CLINICAL TRIAL: NCT06688617
Title: Effect of Swedish Hand Massage on Pain in Patients Undergoing Coronary Artery Bypass Graft Surgery: Randomized Controlled Trial
Brief Title: Effect of Swedish Hand Massage on Pain in Patients Undergoing CABG Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Collaborators: Dr. Siyami Ersek Thoracic and Cardiovascular Surgery Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Oyku Kara, Research Assistant, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 3435-19
Record Dates: First submitted 2024-11-12; First posted 2024-11-14 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Coronary Artery Bypass Graft Surgery (CABG); Pain; Pain Management; Nursing; Massage; Hand Massage
Keywords: Coronary Artery Bypass Graft; Hand Massage; Swedish Massage; Pain; Nursing
MeSH Terms: conditions — Pain; Agnosia

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Swedish hand massage (Experimental): Swedish hand massage was applied to patients who were extubated after the first 4 hours after surgery, were not under the effect of pharmacological or non-pharmacological analgesia, and were in the intensive care period after the first expression of pain.
  Interventions: Other: Swedish Hand Massage
- Control (No Intervention): Patients who were extubated within the first 4 hours after surgery, who were not under the effect of pharmacological or nonpharmacological analgesia, and who were admitted to the intensive care unit with the first pain symptom were followed up during the follow-up periods.

INTERVENTIONS:
Other: Swedish Hand Massage — Swedish technique hand massage: Effleurage-petrissage-friction-tapotement,-vibration-effleurage
  Arms: Swedish hand massage

SUMMARY:
Coronary Artery Bypass Grafting (CABG) surgery is performed commonly today. Heart surgery performed on more than two million individuals every year leads patients experience severe postoperative pain for causes such as cutting of intercostal nerves along the incision line, pleural irritation caused by thoracic catheters etc. Hand massage, which is one of the non-pharmacological methods, is an effective procedure that can be applied independently by nurses for pain management. The objective of this randomized controlled study is to investigate the effect of hand massage applied to the patients with CABG surgery during the postoperative intensive care process, on pain.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent CABG surgery,
* Stated that they were in pain,
* 18 years old and older,
* Had not completed 48 hours after the surgical procedure,
* Accepted to participate in the study verbally and in writing after being informed about the study,
* Could understand the information given,
* Could read, write and speak Turkish,
* Did not have any physiological, psychological or mental problems that would prevent verbal communication,
* Did not have any limb, vascular problem, wound or catheter that would prevent the application of hand massage,
* were ASA classified as I and II,
* Had no previous hand massage experience,
* Did not participate in any other clinical studies during the same period,
* Did not develop any complications during and after the surgical procedure,
* Physiological parameters were within normal limits during the surgical procedure,
* Received the same type of treatment in the post-surgical period,
* Body mass index was within normal limits

Exclusion Criteria:

* Patients who have complications during or after surgical intervention,
* Intubated,
* Have any limb, vascular problem, wound or catheter that prevents hand massage,
* Under the effect of pharmacological or non-pharmacological interventions that will affect pain,
* Obese (body mass index (BMI≥30),

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2018-04-30 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Sternotomy pain | Pain intensity was assessed with a visual analog scale (VAS) before and at 5, 30, 60, 90, 90 and 120 minutes after massage.
Drain pain | Pain intensity was assessed with a visual analog scale (VAS) before and at 5, 30, 60, 90, 90 and 120 minutes after massage.
Back Pain | Pain intensity was assessed with a visual analog scale (VAS) before and at 5, 30, 60, 90, 90 and 120 minutes after massage.
Leg incision pain | Pain intensity was assessed with a visual analog scale (VAS) before and at 5, 30, 60, 90, 90 and 120 minutes after massage.

SECONDARY OUTCOMES:
Systolic blood pressure | Evaluated with a patient monitor before and after the massage at 5, 30, 60, 90, 90 and 120 minutes.
Diastolic blood pressure | Evaluated with a patient monitor before and after the massage at 5, 30, 60, 90, 90 and 120 minutes.
Pulse rate | Evaluated with a patient monitor before and after the massage at 5, 30, 60, 90, 90 and 120 minutes.
Respiratory rate | Evaluated with a patient monitor before and after the massage at 5, 30, 60, 90, 90 and 120 minutes.
Oxygen saturation | Evaluated with a patient monitor before and after the massage at 5, 30, 60, 90, 90 and 120 minutes.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University-Cerrahpaşa, Istanbul, Şişli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
In order to protect the rights of patients, an undertaking was given to the Ethics Committee that the data would not be shared with anyone other than the researchers.